CLINICAL TRIAL: NCT04651335
Title: Comparison of Concentric or Eccentric Virtual Reality Training Program in Subacute-stroke Patients With Hemispatial Neglect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0416
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Neglect
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentric (Active Comparator): uses an afferent virtual reality program
  Interventions: Device: afferent virtual reality program
- Eccentric (Active Comparator): uses an efferent virtual reality program
  Interventions: Device: efferent virtual reality program

INTERVENTIONS:
Device: afferent virtual reality program — When visual gaze training is applied to the left unilateral neglected patient, the gaze direction can be divided into an afferent direction closer to the body and an efferent direction away from the body. The concentric direction moves the ball from the left to the center of the body.
  Arms: Concentric
Device: efferent virtual reality program — When visual gaze training is applied to the left unilateral neglected patient, the gaze direction can be divided into an afferent direction closer to the body and an efferent direction away from the body. The efferent direction moves from the center to the right.
  Arms: Eccentric

SUMMARY:
The purpose of this study is to compare and analyze how the visual gaze training in the afferent direction and the visual gaze training in the efferent direction using virtual reality affects the improvement of the neglect phenomenon in patients with subacute stroke with unilateral neglect.

Based on the behavioral intention test (BIT) test and the Mini-Mental Screening Examination test (MMSE) test for the group of unilateral neglected patients with stroke findings among all eligible patients for this experiment.

Appropriate subjects are selected and randomly divided into two groups. One group uses an afferent virtual reality program, and the other uses an efferent virtual reality program to train five times a week for a total of 4 weeks.

Before training, a computer experience scale 21 was additionally performed, and to find out the degree of unilateral negligence, evaluation was performed using the Behavioral Inattention Test (BIT) and Catherine Bergego Scale (CBS)22, and the angle of deflection (deviation angle), out-of-focus time, gaze time, failure rate, and head rotation trajectory were evaluated. In addition, reaction time, failure rate, and head rotation trajectory were evaluated using a virtual reality program (Assessment program-V2) to evaluate the degree of unilateral negligence. After that, BIT, CBS, and Assessment program-V2 tests are performed to determine the degree of improvement in visual ignorance due to each program.

ELIGIBILITY:
Inclusion Criteria:

1. A person with left hemiplegia who was found to have a stroke by MRI or CT.
2. A person who has been confirmed to have unilateral neglect (BIT 196 or less, or each subtest cut off or less)
3. A person who has enough cognitive ability to receive virtual reality training. (In case of more than 20 points in MMSE)
4. Those within 3 months of onset.

Exclusion Criteria:

1. Those with a history of recurring brain damage
2. hemianopsia
3. When there is a disorder in the movement of the neck due to orthopedic problems
4. Someone has vision and hearing problems during evaluation and treatment
5. difficult to maintain a sitting position in a chair with back and armrests
6. other diseases that may affect your general cognitive decline
7. who disagree with this study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2012-08-09 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Behavioral Inattention Test (BIT) | before treatment
  The Behavioral Inattention Test (BIT) is an objective behavioral test of everyday skills relevant to visual neglect, aimed at increasing the understanding of specific difficulties patients experience.
Behavioral Inattention Test (BIT) | 2weeks
  The Behavioral Inattention Test (BIT) is an objective behavioral test of everyday skills relevant to visual neglect, aimed at increasing the understanding of specific difficulties patients experience.
Behavioral Inattention Test (BIT) | 4weeks
  The Behavioral Inattention Test (BIT) is an objective behavioral test of everyday skills relevant to visual neglect, aimed at increasing the understanding of specific difficulties patients experience.
Behavioral Inattention Test (BIT) | 4weeks after end of the treatment
  The Behavioral Inattention Test (BIT) is an objective behavioral test of everyday skills relevant to visual neglect, aimed at increasing the understanding of specific difficulties patients experience.

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No